CLINICAL TRIAL: NCT01207466
Title: Evaluation of Two Daily Disposable Contact Lenses for Wearers With Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-415-C-001 sub 2
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Astigmatism; Myopia
MeSH Terms: conditions — Astigmatism; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nelfilcon A invest'l / nelfilconA comm'l (Other): Nelfilcon A investigational toric contact lenses worn first, with nelfilcon A commercial toric contact lenses worn second. Each product worn bilaterally on a daily disposable basis for one week.
  Interventions: Device: Nelfilcon A investigational contact lens; Device: Nelfilcon A commercial contact lens
- Nelfilcon A comm'l / nelfilconA invest'l (Other): Nelfilcon A commercial toric contact lenses worn first, with nelfilcon A investigational toric contact lenses worn second. Each product worn bilaterally on a daily disposable basis for one week.
  Interventions: Device: Nelfilcon A investigational contact lens; Device: Nelfilcon A commercial contact lens

INTERVENTIONS:
Device: Nelfilcon A investigational contact lens — Investigational, soft contact lens for astigmatism worn on a daily disposable basis.
Device: Nelfilcon A commercial contact lens — Commercially marketed, soft contact lens for astigmatism worn on a daily disposable basis.
  Other Names: Focus DAILIES Toric

SUMMARY:
The purpose of this trial is to compare the performance of two contact lenses for contact lens wearers with astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing soft contact lenses with astigmatism correction
* Other protocol inclusion criteria may apply

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment
* Currently enrolled in an ophthalmic clinical trial
* Strabismus
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator
* Other protocol exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This reporting group includes all enrolled and dispensed participants. One participant was enrolled but not dispensed due to unacceptable fit. This participant is included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Period: Period 1, One Week of Wear
Arm/Group | Nelfilcon A Invest'l / nelfilconA Comm'l | Nelfilcon A Comm'l / nelfilconA Invest'l
Started | 46 | 48
Completed | 46 (One participant discontinued between Period 1 and Period 2 due to inclusion/exclusion criteria.) | 48
Not Completed | 0 | 0
Period: Period 2, One Week of Wear
Arm/Group | Nelfilcon A Invest'l / nelfilconA Comm'l | Nelfilcon A Comm'l / nelfilconA Invest'l
Started | 45 | 48
Completed | 45 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall
Number analyzed (Participants) | 94
Age Continuous [Mean (Standard Deviation); unit: years] | 35.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Quality of Vision (Crisp and Clear)
Description: Quality of vision (crisp and clear), as interpreted and reported by the participant by eye on a questionnaire as a single, retrospective evaluation of one week's wear time. Quality of vision was assessed on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week of wear
Population: Analysis conducted per protocol, with exclusions due to reasons such as: major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Nelfilcon A Investigational: Investigational, soft contact lenses for astigmatism worn bilaterally on a daily disposable basis for one week.
- Nelfilcon A Commercial: Commercially marketed, soft contact lenses for astigmatism worn bilaterally on a daily disposable basis for one week.
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Number analyzed (Participants) | 92 | 91
Number analyzed (eyes) | 184 | 182
units on a scale | 8.8 (1.3) | 8.6 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 45 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/93
Other Adverse Events (participants affected / at risk) | 0/95 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.